CLINICAL TRIAL: NCT03328273
Title: A Phase 1 Proof-of-Concept Study Investigating AZD6738 Monotherapy and Acalabrutinib in Combination With AZD6738 (ATR Inhibitor) in Subjects With Relapsed or Refractory High-risk Chronic Lymphocytic Leukemia (CLL)
Brief Title: A Study of AZD6738 and Acalabrutinib in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-CL-110; 2016-003737-15 (EudraCT Number); NCT05404282 (obsolete NCT alias)
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ceralasertib; acalabrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A Part 1 and 2 (Other): DISCONTINUED (ceralasertib monotherapy)
  Interventions: Drug: Ceralasertib
- Arm B Part 1 and 2 (Experimental): ceralasertib + acalabrutinib in combination
  Interventions: Drug: Ceralasertib; Drug: Acalabrutinib

INTERVENTIONS:
Drug: Ceralasertib — An ATP competitive, orally bioavailable inhibitor of the Serine/Threonine protein kinase Ataxia Telangiectasia and Rad3 related (ATR).
  Other Names: AZD6738
Drug: Acalabrutinib — An experimental anti-cancer drug and Bruton's tyrosine kinase (BTK) inhibitor.
  Other Names: ACP196
  Arms: Arm B Part 1 and 2

SUMMARY:
This study evaluates the safety, pharmacokinetics, pharmacodynamics and efficacy of acalabrutinib and ceralasertib (known as AZD6738) when taken in combination.

DETAILED DESCRIPTION:
This study is to determine the safety of ceralasertib when given as monotherapy (discontinued) and in combination with acalabrutinib in subjects with R/R CLL and in subjects who have few therapeutic options available to them. As such, this study includes a formal DLT assessment of the first 6-12 subjects dosed in Part 1 of the study. In addition, routine and regular safety monitoring will be undertaken during this study to fully assess safety of ceralasertib given as monotherapy and in combination with acalabrutinib, with toxicity assessment and dose reduction guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed or refractory CLL that meets published diagnostic criteria (International Workshop on Chronic Lymphocytic Leukemia [IWCLL] Hallek 2008) and supported/documented by medical records
* Subjects must be Relapse/Refractory high risk CLL and have exhausted other therapeutic options according to local/regional standard of care
* Must have received ≥1 prior therapy for treatment of their disease.

Exclusion Criteria:

* A diagnosis of ataxia telangiectasia
* Any prior exposure to an ATR inhibitor or known hypersensitivity to an excipient of the product.
* Known history of infection with human immunodeficiency virus (HIV).
* A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ACP-196 (acalabrutinib) and/or Ceralasertib
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or corrected QT interval (QTc) > 480 msec.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* Requirement of treatment with proton-pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Subjects receiving proton-pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
* Breast feeding or pregnant

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing dose-limiting toxicities | 28 Days
  Arm A (discontinued): When given as monotherapy in subjects with R/R high-risk CLL who have exhausted other therapeutic options according to local/regional standard of care.
  Arm B: Ceralasertib given in combination with acalabrutinib in subjects with R/R high-risk CLL who are suitable for treatment with a BTK inhibitor and ceralasertib, per investigator's clinical opinion.

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613; acertamc@dlss.com
Locations (10):
- Poland (2):
  - Research Site, Krakow
  - Research Site, Lodz
- United Kingdom (8):
  - Research Site, Birmingham
  - Research Site, Bournemouth
  - Research Site, Cardiff
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Oxford
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Jurczak W, Elmusharaf N, Fox CP, Townsend W, Paulovich AG, Whiteaker JR, Krantz F, Wun CC, Parr G, Sharma S, Munugalavadla V, Manwani R, Dean E, Munir T. Phase I/II results of ceralasertib as monotherapy or in combination with acalabrutinib in high-risk relapsed/refractory chronic lymphocytic leukemia. Ther Adv Hematol. 2023 May 30;14:20406207231173489. doi: 10.1177/20406207231173489. eCollection 2023. PMID 37273420
- See also: redacted_CSR_synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-110&attachmentIdentifier=8cd9b89c-d75b-4b6e-8b0b-ac9b4ff4e6ba&fileName=D5330C00008abbreviatedCSRsynopsis_redacted_Final_26Jan2022.pdf&versionIdentifier=